CLINICAL TRIAL: NCT04468906
Title: Tenodesis vs. Self-locking Tenotomy in Long Head of the Biceps Tendon Lesions: A Randomized Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was closed due to difficulty in recruitment of target population.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-01026
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Tenodesis; Tenotomy
Keywords: LHBT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biceps self-locking "T" tenotomy (Experimental)
  Interventions: Procedure: Self-locking "T" Tenotomy
- Biceps tenodesis (control) (Active Comparator)
  Interventions: Procedure: Biceps Tenodesis

INTERVENTIONS:
Procedure: Biceps Tenodesis — Biceps tenodesis describes the surgical procedure that will be performed to treat LHBT lesions.
  Arms: Biceps tenodesis (control)
Procedure: Self-locking "T" Tenotomy — Self-locking "T" Tenotomy describes the surgical procedure that will be performed to treat LHBT lesions.
  Arms: Biceps self-locking "T" tenotomy

SUMMARY:
One of the common complaints after long head of the biceps brachii tendon (LHBT) surgery is a Popeye deformity, which can occur with both the tenodesis and tenotomy. Tenotomy using the traditional technique has a higher incidence of Popeye deformity as the residual stump is not fixated in place. However, the more recently-described self-locking tenotomy improves upon this by having a wider stump base to theoretically prevent reduce the incidence of tendon retraction down the bicipital groove. If this technique is shown to result in a similar incidence of Popeye deformity, then it may be preferable to tenodesis due to its advantages of reduced postoperative pain, more rapid return to activity, and reduced surgical time and cost. The purpose of the proposed study is to evaluate the effect of biceps tenodesis versus self-locking T tenotomy in the management of lesions involving the LHBT.

DETAILED DESCRIPTION:
Long head of the biceps brachii tendon (LHBT) lesions are a common pathology and can be a significant source of pain in the shoulder due to the large number of free nerve endings around the tendon. There are 3 main subtypes of LHBT lesions 1) LHBT degeneration, 2) LHBT anchor disorders, and 3) LHBT instability. These lesions can occur both in isolation or in conjunction with rotator cuff disease. Treatment options include tenotomy and tenodesis, and while both are utilized there exists a lack of consensus treatment choice.

The optimal management of LHBT lesions remains controversial, with surgeons typically treating younger patients with tenodesis and older patients with tenotomy. Previous RCTs have failed to discern a clinical difference between tenodesis and tenotomy, apart from the reduced incidence of Popeye deformity in the tenodesis cohorts. However, all previous literature has utilized the traditional biceps tenotomy technique of transecting the tendon just lateral to its insertion on the superior labrum. This results in a narrow tendon stump that usually slips through the transverse humeral ligament and retracts down the arm, resulting in the aforementioned deformity. A newer tenotomy technique, termed the self-locking tenotomy, consists of preserving the attachment of the LHBT on the superior labrum and instead releasing the superior labrum off the glenoid from the 11 o'clock to 1 o'clock positions. As a result, the residual LHBT stump is broad and "T-shaped", which has a lower incidence of retracting down the arm. Using this technique, LHBT tenotomy has been shown to result in similar rates of Popeye deformity as the tenodesis in a number of recent case series.

This will be a single-center randomized controlled trial. The study is comparing biceps tenodesis and self-locking tenotomy in patients undergoing arthroscopic shoulder surgery for lesions involving the LHBT.

ELIGIBILITY:
Inclusion Criteria:

* Primary indication is for pathology of the LHBT or biceps-labrum complex
* Age 40-80
* Ability to comply with a standardized postoperative protocol
* Willing and able to provide consent

Exclusion Criteria:

* Associated rotator cuff tear requiring arthroscopic repair
* Pregnant patient
* Age <40 years
* Previous shoulder surgery
* Unable to speak English or perform informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Rate of Reverse Popeye Deformity | up to 24 months post-op
  Reverse popeye deformity is the loss of the theoretical LHBT stabilizing effect on the humeral head, which can be determined with a physical exam.

SECONDARY OUTCOMES:
Change in Score on American Shoulder & Elbow Surgeons (ASES) Scale | 6 months post-op, 24 months post-op
  The ASES scale consists of two subscales: pain (0-50 points) and function/disability (0-50 points), with a total score range of 0-100 points. The lower the score, the greater the pain and disability.
Change in Score on Visual Analogue Scale (VAS) | 6 months post-op, 24 months post-op
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain possible." The total score range is 0-10. The higher the score, the higher the pain level experienced.
Incidence of fatigue, cramping, biceps groove tenderness | up to 24 months post-op
Average timing of return to work/sport | up to 24 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Laith Jazrawi, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to use the data upon reasonable request. Requests should be directed to laith.jazrawi@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.